CLINICAL TRIAL: NCT07006675
Title: Effect of NSAIDs on Union, Opioid Utilization and Pain Management for Tibia Fractures: A Pragmatic, Randomized Controlled Trial
Acronym: NSAID
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Major Extremity Trauma Research Consortium (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: W81XWH-15-2-0058
Record Dates: First submitted 2025-05-27; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Tibial Fractures; Pain
Keywords: Ibuprofen; Pain Management; Tibia Fracture; IM Nail Fixation; NSAID
MeSH Terms: conditions — Tibial Fractures; Pain; Agnosia | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care Pain Management with NSAIDs (Active Comparator): Treatment patients will receive oral ibuprofen 600 mg three times a day (tid) for up to six weeks. Clinicians in this group may use whatever further analgesia they desire, excluding NSAIDs. For patients who have a clinical concern regarding NSAID and prophylactic anticoagulation, the treating physician may consider prescribing misoprostol.
  Interventions: Drug: 600 mg Ibuprofen
- Standard of Care Pain Management without NSAIDs (No Intervention): Control patients will receive standard of care pain medication regimen and may not use NSAIDs. Clinicians in this group may use whatever further analgesia they desire, excluding NSAIDs.

INTERVENTIONS:
Drug: 600 mg Ibuprofen — Treatment patients will receive oral ibuprofen 600 mg three times a day (tid) for up to six weeks. Clinicians in this group may use whatever further analgesia they desire, excluding NSAIDs. For patients who have a clinical concern regarding NSAID and prophylactic anticoagulation, the treating physician may consider prescribing misoprostol.
  Other Names: Advil; Motrin
  Arms: Standard of Care Pain Management with NSAIDs

SUMMARY:
Two arm, pragmatic, randomized controlled multicenter Phase III noninferiority trial evaluating the efficacy of standard pain management without NSAIDs (Group 1) vs. standard pain management plus up to 6 weeks of NSAIDs (Group 2) in the treatment of tibial shaft fractures.

DETAILED DESCRIPTION:
The proposed study is a two arm, pragmatic, randomized controlled multicenter Phase III noninferiority trial. We will randomize patients with diaphyseal tibia fractures treated with intramedullary (IM) nail into two treatment arms. The control group will receive standard pain management with no NSAIDs. The treatment intervention group will receive standard pain management plus up to six weeks of NSAIDs (3 weeks of prescribed medication followed by 3 weeks of medication PRN). Our hypothesis is that pain management using up to 6 weeks of NSAIDs will result in improved pain control and lower opioid consumption but demonstrate non-inferior levels of complications compared to standard of care pain management. The aim of the study is to:

Specific Aim: Evaluate the effect of standard pain management without NSAIDs (Group 1) vs. standard pain management plus up to 6 weeks of NSAIDs (Group 2) in the treatment of tibial shaft fractures.

Primary Hypothesis: When compared to patients who received standard of care pain management, patients treated with up to 6 weeks of NSAIDs will have noninferior rates of surgery for nonunion at one year.

Secondary Hypotheses: When compared to patients who received standard of care pain management without NSAIDs, patients treated with up to 6 weeks of NSAIDs will benefit from (1) reduced opioid utilization; (2) reduced levels of persistent pain; (3) reduced pain interference; (4) improved functional outcomes; (5) noninferior rates of analgesic treatment related side effects; and (6) noninferior rates of radiographic union.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with open (Grade I, II, of IIIa) or closed tibia fractures treated with a nail.
2. Patients 18-80 years old inclusive.
3. Patients able to be followed at a METRC facility for at least 12 months following injury

Exclusion Criteria:

1. Patient unable to provide informed consent
2. Patients who are current - intravenous drug user.
3. Patients with a history of allergy to the study drugs.
4. Patients unable to swallow oral medications or without functioning GI tract.
5. Patients with a history of gastrointestinal bleeds or gastric perforation.
6. Patients with a history of stroke or heart attack.
7. Patients requiring an aspirin or NSAID regimen except for low dose aspirin, 81mg.
8. Patients with any bleeding disorders.
9. Patients with severe renal failure [GFR:<30]. Patients with moderate renal failure [GFR: 30-59] may participate in the study at a modified dose [see section 8.6 for defined modified dose].
10. Patients undergoing daily treatment with systemic glucocorticoids before surgery.
11. Patients likely to have severe problems maintaining follow-up, including patients diagnosed with a severe psychiatric conditions, patients who live too far outside the hospital's catchment area, patients who are incarcerated and patients who have unstable housing situations.
12. Patients with a GCS <15 at discharge.
13. Patients with a closed head injury that precludes NSAIDS.
14. Patients who are pregnant or lactating at time of screening
15. Patients with a bone graft procedure planned for a future date at the time of initial definitive fixation surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Secondary surgery to promote bone union after 3 months post initial surgery | 1 year
  Bone nonunion will be assessed by the presence of a secondary surgery to promote union after 3 months and up to 12 months post definitive fixation surgery. Non-prophylactic secondary surgery to promote union will be considered evidence of nonunion. Each case will be independently reviewed by members of the METRC Central Adjudication Committee and if at least 2 members agree with the assessment of secondary surgery to promote union, no further review will be necessary. The METRC Central Adjudication Committee will convene to discuss the cases for which there is disagreement regarding non-union assessment.

SECONDARY OUTCOMES:
Opioid Utilization | 1 year
  Opioid utilization will be recorded in two ways: Opiate pain medicine prescribed by the treating provider as well as self -reported opiate use by the study subjects.
Adverse Effects and Complications | 1 year
  Adverse effects and complications of ibuprofen include, in addition to nonunion, wound closure complications, bleeding complications, as well as pain treatment related adverse effects. Adverse effects include nausea, vomiting, dizziness, headaches, renal impairment, platelet inhibition and angioedema. In addition, on 7/9/15 the FDA released an announcement related to the risks of NSAIDS entitled, "FDA Drug Safety Communication: FDA strengthens warning that non-aspirin non-steroidal anti-inflammatory drugs (NSAIDs) can cause heart attacks or strokes". 45 Consequently, consent forms for this study will include the required language and participants will be assessed for these cardiovascular outcomes.
Persistent Pain & Pain Inference | 1 year
  The BPI (Brief Pain Inventory) is a widely used, 15-item measure of pain intensity and interference with daily life and will be assessed at baseline, 3, 6, and 12 months post definitive fixation surgery. It has been extensively validated in both English and Spanish, and also includes questions about pain treatments and the effectiveness of these treatments.46 The BPI pain intensity domain is compatible with the IMMPACT guidelines for assessing pain in clinical trials and the FDA Guidance for Industry on the use of Patient-Reported Outcome Measures. In addition to the BPI instrument, pain inference will be collected using the Patient Report Outcomes Measurement Information System (PROMIS) as described below.
Physical and Psychosocial Function | 1 year
  Self -Reported Measures of Physical and Psychosocial Function will be assessed at baseline, 3, 6, and 12 months post definitive fixation surgery using the Patient Report Outcomes Measurement Information System (PROMIS) Computer Adaptive Test (CAT) item banks, a product of the NIH Roadmap for Medical Research. CATs present an advantage over traditional measures in that they target only the most relevant items to each patient and can thus be used to obtain precise measurements with 4-6 items, making assessment across multiple domains feasible. CATs can also extend the ceiling and floor of individual domains, potentially enhancing responsiveness. At any visit if a CAT cannot be administered, respondents will instead complete the appropriate short forms associated with the CAT measure.
Radiographic bone union | 1 year
  Radiographic union will be based on the modified RUST score44 assessed between 3 months and 12 months after definitive fixation surgery. Radiographic examinations at 3, 6 and 12 months by an adjudication committee comprised of METRC investigators will be evaluated based on AP and lateral x-rays.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Higgins, MD, Principal Investigator — University of Utah; Renan Castillo, PhD, Principal Investigator — Johns Hopkins University
Locations (14):
- United States (13):
  - Eskenazi Hospital, Indianapolis, Indiana
  - Indiana University-Methodist, Indianapolis, Indiana
  - University of Maryland R Adams Cowley Shock Trauma Center, Baltimore, Maryland
  - Harvard Medical Center, Cambridge, Massachusetts
  - Hennepin Health, Minneapolis, Minnesota
  - University of Mississippi, Jackson, Mississippi
  - The MetroHealth System, Cleveland, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Vanderbilt Medical Center, Nashville, Tennessee
  - University of Texas Health Science Center - Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Inova Fairfax Hospital, Falls Church, Virginia
  - University of Wisconsin, Madison, Wisconsin
- University of Calgary, Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided